CLINICAL TRIAL: NCT02153229
Title: A Randomized Phase 2 Trial of Radical Pleurectomy and Post-Operative Chemotherapy With or Without Intraoperative Porfimer Sodium -Mediated Photodynamic Therapy for Patients With Epitheliod Malignant Pleural Mesothelioma
Brief Title: Phase II Trial of Radical Pleurectomy With or Without Intraoperative PDT for Malignant Pleural Mesothelioma
Acronym: MPM-PDT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 14513
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Epitheliod Malignant Pleural Mesothelioma
Keywords: Histological diagnosis of MPM; epitheliod subtype; limited to the hemithorax; macroscopically complete resection of the tumor
MeSH Terms: interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Drug Therapy; Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- patients who undergo RP plus photofrin-based PDT (Experimental)
  Interventions: Radiation: Photodynamic Therapy; Procedure: Radical Pleurectomy; Radiation: Chemotherapy; Drug: Photofrin 2.0 mg/kg
- patients who undergo RP alone (Experimental)
  Interventions: Procedure: Radical Pleurectomy; Radiation: Chemotherapy

INTERVENTIONS:
Radiation: Photodynamic Therapy
  Other Names: PDT
  Arms: patients who undergo RP plus photofrin-based PDT
Procedure: Radical Pleurectomy
  Other Names: RP
Radiation: Chemotherapy
Drug: Photofrin 2.0 mg/kg — If randomized to the RP with PDT arm, subject will receive Photofrin 2.0 mg/kg as an intravenous infusion 24 hours (range 18-30 hours) prior to intra-operative light delivery (PDT) during radical pleurectectomy
  Arms: patients who undergo RP plus photofrin-based PDT

SUMMARY:
A randomized Phase II trial to test whether the addition of intraoperative Photofrin-mediated photodynamic therapy to radical pleurectomy and post-operative chemo.improves OS in the treatment of patients with epithelioid MPM. Subjects assigned to the PDT arm will be given the photosensitizer prior to surgery . All subjects will receive maximal surgical debulking. Subjects in the PDT arm will receive intraoperative treatment using real-time, isotropic light dosimetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of MPM, epithelioid subtype, who in the opinion of the attending thoracic surgeon can receive a macroscopically complete resection of tumor.
* Patients must have disease limited to the hemithorax.
* Patients who have received prior surgery, gene therapy, or combination chemotherapy will be permitted if it has been at least 30 days since the last treatment.
* Subjects treated with pemetrexed previously will be eligible only if 30 days have elapsed between the last dose of pemetrexed and the date of surgery.
* ECOG performance status of 0-1.
* Medical suitability for resection, including documented medical and cardiac clearance.
* 18 years of age or older.
* Patients must sign a document that indicates that they are aware of the investigative nature of the treatment of this protocol, and the potential benefits and risks. Patients unwilling or unable due to cognitive impairment to sign informed consent are excluded from the study.

EXCLUSION CRITERIA

* Patients with active invasive cancers, other than MPM, that require additional treatment, except non-melanomatous skin cancer, superficial bladder or cervical cancer, and early-stage prostate cancer
* Pregnant or lactating patients.
* Patients who have a history of HIV disease.
* Patients who have a white count less than 2,500 per cubic mm or platelets less than 100,000/cubic mm.
* Serum creatinine equal or greater than 2.5 mg/deciliter.
* Patients who have severe liver disease including cirrhosis, Grade III-IV elevations in liver function studies, or bilirubin in excess of 1.5 mg/deciliter.
* Patients with porphyria or hypersensitivity to porphyrin or porphyrin-like compounds.
* Patients who have been treated with pemetrexed if the last dose of pemetrexed is < 30 days to the date of surgery.
* Patients that have been treated with prior Mantle field radiation.
* Patients with distant metastatic disease or otherwise not confined to the ipsilateral hemithorax.
* Subjects who have received more than 2 doses of neo-adjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival months | 4 years

SECONDARY OUTCOMES:
Progression-free survival months | 4 years
Local Control | 4 years
  progression with death as a competing risk
Receipt of Pembrolizumab | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania